CLINICAL TRIAL: NCT05936164
Title: The Nigeria National Registry of Atrial Fibrillation
Brief Title: Nigeria Atrial Fibrillation Registry
Acronym: NigAfibReg
Status: Not yet recruiting | Type: Observational
Sponsor: University College Hospital, Ibadan (Other)
Responsible Party: Principal Investigator, O.S Ogah, DR, University College Hospital, Ibadan
Other Study IDs: NigAfibRegistry_V.2
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation, arrhythmias, heart failure
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial fibrillation is the most common sustained cardiac arrhythmia (rhythm abnormality) encountered in clinical practice. It contributes significantly to the risk of cardiac symptoms, hospital admissions, cardiovascular related morbidity and mortality and increased healthcare cost.

AF has significant impact on healthcare cost. The major drivers of the cost are hospitalisations, stroke and loss of productivity. Globally AF accounts for less than 1% of all deaths. However, because it co-exists with other conditions, it contributes to worse prognosis compared to persons who do not have AF. New onset AF in HF patients may be associated with particularly poor prognosis.

Most of the published data and current knowledge on AF epidemiology are based on studies in Europe and North America. The information obtainable from previous studies in sub-Saharan Africa is limited. Many of the studies were retrospective. There is also paucity of information on burden of AF (both in hospital and community), clinical profile and outcome of AF in Nigeria in particular and Africa in general.

The primary objective of this study is to determine the clinical characteristics, outcome as well as cost genetic features of AF in Nigeria.

The project will provide information on: i. Hospital and community burden of AF in Nigeria; ii. Clinical features, mode of presentation and risk factors for AF; iii. Provide data on AF related outcomes as well as prognostic factors.

DETAILED DESCRIPTION:
Background to the Research Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia (rhythm abnormality) encountered in clinical practice. (1) It contributes significantly to the risk of cardiac symptoms, hospital admissions, cardiovascular related morbidity and mortality and increased healthcare cost. (1, 2) In 2010, the Global Burden of Disease (GBD) study estimated that about 33.5 million people have AF globally which represents about 0.5% of the world population. (2) The increasing rate of AF has been attributed to the ageing of the world population, rise in the burden of cardiovascular risk factors such as overweight/obesity, high blood pressure, diabetes mellitus etc. (1, 2) In 2010, the Global Burden of Disease (GBD) study estimated that about 33.5 million people have AF globally. Between 1990 and 2010, the total number of deaths associated with AF in sub-Saharan Africa (SSA) increased from 441 to 1227 (196% change) The age standardized death rate (per 100,00) associated with AF rose from 0.4 to 0.6 (50% change) between 1990 and 2013. (1) Nigeria contributes to a large proportion of AF in SSA and little attention has been paid to this huge health problem.

Statement of the Problem AF has been shown to be associated with increased morbidity (especially increased association with the risk of development of heart failure (HF) and stroke, in addition to increased risk of mortality. AF is also a significant public health problem based on the fact that it accounts for about 1% of the National Health Service budget in many countries. In the United States of America (USA), the management of AF consumes about 16-26 billion dollars annually. The recent global burden of disease report has provided evidence of progressive increases in the overall burden, incidence, prevalence as well as AF associated mortality in ten-year period (1990-2010) in Africa and Nigeria contributes to a large proportion of this. Aging of the population is associated with vascular disease due to hypertension, atherosclerosis and other CVD risk factors which increase arterial stiffness, cause diastolic dysfunction and atrial volume overload resulting in AF. Most of the published data and current knowledge on AF epidemiology are based on studies in Europe and North America. The information obtainable from previous studies in sub-Saharan Africa is limited. Many of the studies were retrospective. There is also paucity of information on burden of AF (both in hospital and community), clinical profile and outcome of AF in Nigeria in particular and Africa in general.

Objectives of the Research Primary Objective The primary objective of this study is to determine the clinical characteristics, outcome as well as cost genetic features of AF in Nigeria.

Secondary Objectives-

1. To determine the hospital prevalence, clinical features and modes of presentation of AF in Nigeria.
2. To conduct and determine the community prevalence of AF in Nigeria
3. To determine the risk factors of AF in Nigeria.
4. To determine the complications of AF in Nigeria
5. To ascertain the mode of management of AF in Nigeria.
6. To determine the 12-months outcome of the condition and develop predictive models of outcome for AF in the country.

Research Questions

1. What are the hospital and community prevalence of AF in Nigeria.
2. What are the clinical features and modes of presentation of AF in Nigeria?
3. What are the risk factors of AF in Nigeria?
4. What are the complications of AF in Nigeria?
5. What are the modes of management of AF in Nigeria?
6. What are the 12-months outcomes of AF in the country and are there predictive models of outcome in the country? Brief Literature Review Globally it is estimated that there 2.7 million new cases in males and 2.0 million cases in females of AF. (1) The age adjusted mortality rate 1.6 and 1.7 for men and women respectively of AF has been reported. In terms of disability adjusted life years (DALYs), this is estimated as 64.5 and 45.9 per 100,000 populations for men and women respectively. (1) AF is associated with increased risk of mortality after adjusting for other confounders. In the Framingham Heart Study, AF was associated with 1.5-1.9-fold increase in mortality in over 40-years of follow-up. In the Olmsted County Study, the mortality associated with AF at 4- and 12- months was 17 and 23% respectively. Elderly individuals (aged 70 years and above in rural Tanzania have 1-year mortality of 50% and 66.6% in men and women respectively AF has significant impact on healthcare cost. The major drivers of the cost are hospitalisations, stroke and loss of productivity (3) Globally AF accounts for less than 1% of all deaths. However, because it co-exist with other conditions, it contributes to worse prognosis compared to persons who do not have AF. New onset AF in HF patients may be associated with particularly poor prognosis. (3) There is limited data on population/ hospital prevalence and incidence of AF in SSA in general and Nigeria (Africa's most populous nation in particular) The very few hospitals based data are from Cameroon, Ivory Coast, Kenya, Senegal and South Africa. Most were retrospective report. The few from Nigeria recruited very few subjects (less than 100) (4) In South Africa about 4.6% of patients seen in a cardiac clinic had AF giving a prevalence of 5.6/100,000 population per year. (16) The estimated prevalence in Ivory Coast is 5.5/100,000 population based on a retrospective review over a 10-year period. AF prevalence in Senegal was estimated as 5.4% and it accounted for 66% of all heart rhythm disorders in the country. About 162 patients out of 22,144 medical patients were reported to have AF /Flutter in a private tertiary hospital in Kenya giving a prevalence of 0.7%.

In a community-based study in Tanzania, the crude prevalence of AF was low (0.7%). This is lower than similar study in Europe and North America where the prevalence is about 10% (in those aged 80 years and above) and 5% in those aged 65 years and above respectively.

The prevalence of AF among Africa Americans is strikingly lower compared to their Caucasian counterpart even when the risk factors for AF are higher in the former.

Research Methodology Design The study shall be prospective, observational and shall be conducted in 6 hospitals in the six geopolitical regions of the country. The community survey shall be cross-sectional in randomly selected urban and rural areas in the six geopolitical regions in the country Study population Subjects are eligible to participate if they are 18 years and above and have 12-lead ECG features of AF.

Exclusion criteria Subjects who refuse to participate in the study and pregnant women. Consent Written and/or informed consent shall be obtained from the subjects prior to enrolment into the study.

Enrollment and data collection All subjects with clinical diagnosis of AF shall be recruited. Data from each subject shall be obtained using a uniform and standardized case report forms and a detailed clinical documentation on newly diagnosed/ newly presenting cases/ pre-existing cases of HF shall be carried out. The following data shall be obtained: study identification number, centre code, demographic data, date of diagnosis of HF and pre-admission history (previous heart failure related admissions). Others include NYHA functional class, symptoms, signs, self-reported cardiovascular risk factors, aetiological risk factors/ co-morbidities, blood investigations, 12-lead ECG, echocardiography, medications and 12-month outcome.

Follow up Follow-up of subjects shall be through clinic visits or via telephone (if patient can't come to the clinic). Telephone numbers of next of kin of patients shall also be obtained. The follow up period shall be at one month, six month and 12 months from the time of consent. This will be conducted through the use of research nurses. Information that shall be obtained during the follow-up period includes well-being of the patient, symptoms, signs, medications as well as outcome.

Data analysis Data shall be entered by experienced personnel on personal computers and analyzed with SPSS version 11.0 (SPSS, Inc. Chicago Illinois) Other statistical packages such as STATA and SAS shall be used where necessary. Descriptive statistics for baseline data will be performed on continuous variables using mean, standard deviation, range and median where appropriate. Categorical variables shall be expressed as percentages. McNemar and chi-square tests (for categorical variables) and Student's t-test or analysis of variance (for continuous variables) shall be used for comparisons as appropriate. Advanced statistical analysis e.g. regression analysis shall be applied as necessary.

Data dissemination plan Publication policy will be decided by a writing committee consisting of all the members of the steering committee and the principal investigators from all participating sites. However, all the members of the steering committee, all principal investigators and all those considered by the steering committee to have contributed sufficiently to the study will be co-authors of the primary publications.

Expected Results The project will provide information on: i. Burden of AF in Nigeria; ii. Clinical features, mode of presentation and risk factors for AF; iii. Provide data on AF related outcomes as well as prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

All cases of confirmed atrial fibrillation

Exclusion Criteria:

Refusal of consent

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects are eligible to participate if they are 15 years and above and have 12-lead ECG features of atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 12 months
  All deaths

SECONDARY OUTCOMES:
Hospitalisation | At 12 months
  All hospital readmissions
Stroke | 12 months
  All forms of stroke
Any other thromboembolic events | 12 months
  Any other thromboembolic events